CLINICAL TRIAL: NCT04679168
Title: Change of Environmental Chemical Exposures and Prevalence of Chronic Kidney Disease After Epidemiological Spread of SARS-CoV-2 (COVID-19)
Brief Title: Study on Kidney Disease and EnviromenTal Chemical
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung Pyo Lee, Principal Investigator, M.D., Ph.D., Seoul National University Hospital
Other Study IDs: SKETCH
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Environmental Exposure; Chronic Kidney Diseases
Keywords: COVID-19; Environmental Exposure; Behavioral changes; Chronic kidney disease
MeSH Terms: conditions — COVID-19; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — * Method of obtaining human-derived material samples: Acquiring about 10 ml of urine and 1 ml or more and less than 2 ml of serum samples
  * For blood (serum) samples, residual samples after the tests performed for the clinic visit are used, and urine samples are newly collected at the clinic visit
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Purpose: To confirm the changes in lifestyle due to differences in perceptions of infectious disease risk after the COVID-19 pandemic, decrease in exposure levels of environmentally hazardous chemicals and changes in indicators related to chronic kidney disease
2. Methods:

   * Survey on health risk awareness and lifestyle for COVID-19
   * Blood and urine tests for exposure to environmentally hazardous chemicals
   * Collection of hospital clinical data utilization for indicators related to chronic kidney disease
3. Clinical endpoints:

   * Verification of differences in health risk perception level and lifestyle changes
   * Verification of changes in lifestyle changes and exposure to environmentally hazardous chemicals
   * Verification of changes in indicators related to kidney disease according to changes in exposure to environmentally hazardous chemicals
4. Statistical methods: chi-square test, independent mean comparison t-test, ANOVA test, regression analysis

DETAILED DESCRIPTION:
1. Background In daily life, people are exposed to various environmental hormones (Endocrine Disrupting Chemicals) such as phthalates, bisphenols, heavy metals, and perfluorinated compounds. Due to the recent pandemic of the COVID-19, behavior patterns such as wearing a mask and refraining from going out in daily life have changed. Such behavioral changes have the potential to change the level of exposure to environmental hazards, like intervention studies. In addition, studies have been reported that exposure to various environmental hormones can affect kidney function, but epidemiological studies are insufficient. Therefore, the research team is trying to determine whether exposure to environmental hormones changes due to changes in behavioral patterns according to the new corona epidemic, and to determine the effect on renal function indices in patients with chronic kidney disease.
2. Hypothesis and Purpose

   * Differences in risk perception for disease after the COVID-19 pandemic can explain the degree of change in lifestyle.
   * The changed lifestyle will lead to reduced exposure to environmentally hazardous substances.
   * Reduction of exposure to environmentally harmful substances will reduce the level of exposure to harmful substances related to kidney disease, which will lead to changes in the prevalence of kidney disease and indicators related to kidney disease.
   * After the COVID-19 pandemic, it is verified whether the exposure level of environmentally hazardous chemicals decreases due to changes in the way of life and differences in perception of the risk of infectious diseases, and confirms which indicators related to chronic kidney disease change accordingly. Identify the role.
3. Methods (1) During the COVID-19 pandemic

   * Acquisition of consent (using explanations and posters) by explaining the research purpose and method
   * Survey on changes in awareness of diseases and changes in hygiene activities since the COVID-19 pandemic compared to before
   * Measurement of the concentration of environmentally hazardous substances through the acquisition of blood (serum, residual samples after blood tests for treatment) and urine samples that are normally performed in the office (3 months cycle, 4 times)
   * Acquisition of clinical information related to kidney disease (2) Recovery period of the COVID-19 pandemic
   * Survey on changes in awareness of diseases and hygiene activities that have changed since the end of the COVID-19 outbreak
   * Measurement of the concentration of environmentally harmful substances by obtaining blood (serum, residual sample after blood test for medical treatment) and urine sample (once after 6 months of termination)
   * Acquisition of clinical information related to kidney disease (3) Investigation variable

     a) Survey
   * Demographic information
   * Anthropometric information
   * Risk perception for the COVID-19
   * Individual behavior associated with hygiene
   * Social distancing pattern b) Chemical material in human sample (blood, urine)
   * Phthalate metabolite
   * Paraben metabolite
   * Benzophenone
   * Triclosan and triclocarban
   * Bisphenols
   * Phosphate metabolites
   * Organochlorine pesticides
   * Polychlorinated biphenyls c) Clinical information including estimated glomerular filtration rate, urine protein/creatinine ratio

ELIGIBILITY:
Inclusion Criteria:

* aged 19 years or older
* who have been treated twice or more with chronic kidney disease as their main diagnosis in an outpatient department of kidney medicine for more than 3 months

Exclusion Criteria:

* Patients who do not observe the rapid deterioration of renal function (AKI)
* Patients who are likely to significantly change their lifestyle and exposure levels of environmentally hazardous chemicals due to the rapid progression of the disease itself, accompanied by the following chronic diseases (malignant tumors, dementia, immunosuppressants Use, stroke within 1 year, cerebral hemorrhage, myocardial infarction)
* Other patients who have difficulty in general communication or who are unable to carry out their daily life on their own

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Target number: around 310
  * The total number of participants in the study is around 300-350. In order to figure outcomes, data from the Basic Survey on National Environmental Health were used, and the preceding study (intervention study) was referred to.
  * In multiple regression analysis, the correlation between eGFR and ethylparaben (EtP) was examined by adjusting age, BMI, smoking history, and drinking history. In the full model, where all variables were corrected, R2 was 0.478, and when the independent variable EtP was excluded, R2 decreased by 0.012. Based on these values, as a result of setting the power of 0.7, 0.8, and 0.9 in the multiple regression model, n = 283, 359, and 479, respectively. Based on this result, the number of study participants was set to around 300-350.
Sampling Method: Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of environmental hazard exposure levels and influencing factors | From initial recruitment to after 21 (+/- 3) months
  * Collecting and organizing survey data
  * Calculation of technical statistics on exposure to major environmental hazards
  * Identification of determinants affecting the exposure level of environmentally hazardous substances
Relationship between exposure and health related behavior change | From initial recruitment to after 21 (+/- 3) months
  * Analysis of correlation of kidney disease occurrence according to exposure to harmful substances
  * Identify the possibility of health effects from exposure to environmentally harmful factors such as disease prevalence, glomerular filtration rate, and urine protein/creatinine ratio according to the definition of chronic kidney disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Pyo Lee, M.D., Ph.D., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul National University Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Street ME, Angelini S, Bernasconi S, Burgio E, Cassio A, Catellani C, Cirillo F, Deodati A, Fabbrizi E, Fanos V, Gargano G, Grossi E, Iughetti L, Lazzeroni P, Mantovani A, Migliore L, Palanza P, Panzica G, Papini AM, Parmigiani S, Predieri B, Sartori C, Tridenti G, Amarri S. Current Knowledge on Endocrine Disrupting Chemicals (EDCs) from Animal Biology to Humans, from Pregnancy to Adulthood: Highlights from a National Italian Meeting. Int J Mol Sci. 2018 Jun 2;19(6):1647. doi: 10.3390/ijms19061647. PMID 29865233
- [Background] Grandjean P, Bellanger M. Calculation of the disease burden associated with environmental chemical exposures: application of toxicological information in health economic estimation. Environ Health. 2017 Dec 5;16(1):123. doi: 10.1186/s12940-017-0340-3. PMID 29202828
- [Background] Mascarelli A. Environment: toxic effects. Nature. 2012 Mar 15;483(7389):363-5. doi: 10.1038/nj7389-363a. No abstract available. PMID 22432121
- [Background] Watts N, Amann M, Ayeb-Karlsson S, Belesova K, Bouley T, Boykoff M, Byass P, Cai W, Campbell-Lendrum D, Chambers J, Cox PM, Daly M, Dasandi N, Davies M, Depledge M, Depoux A, Dominguez-Salas P, Drummond P, Ekins P, Flahault A, Frumkin H, Georgeson L, Ghanei M, Grace D, Graham H, Grojsman R, Haines A, Hamilton I, Hartinger S, Johnson A, Kelman I, Kiesewetter G, Kniveton D, Liang L, Lott M, Lowe R, Mace G, Odhiambo Sewe M, Maslin M, Mikhaylov S, Milner J, Latifi AM, Moradi-Lakeh M, Morrissey K, Murray K, Neville T, Nilsson M, Oreszczyn T, Owfi F, Pencheon D, Pye S, Rabbaniha M, Robinson E, Rocklov J, Schutte S, Shumake-Guillemot J, Steinbach R, Tabatabaei M, Wheeler N, Wilkinson P, Gong P, Montgomery H, Costello A. The Lancet Countdown on health and climate change: from 25 years of inaction to a global transformation for public health. Lancet. 2018 Feb 10;391(10120):581-630. doi: 10.1016/S0140-6736(17)32464-9. Epub 2017 Oct 30. No abstract available. PMID 29096948
- [Background] Obrador GT, Schultheiss UT, Kretzler M, Langham RG, Nangaku M, Pecoits-Filho R, Pollock C, Rossert J, Correa-Rotter R, Stenvinkel P, Walker R, Yang CW, Fox CS, Kottgen A. Genetic and environmental risk factors for chronic kidney disease. Kidney Int Suppl (2011). 2017 Oct;7(2):88-106. doi: 10.1016/j.kisu.2017.07.004. Epub 2017 Sep 20. PMID 30675423
- [Background] Song JY, Yun JG, Noh JY, Cheong HJ, Kim WJ. Covid-19 in South Korea - Challenges of Subclinical Manifestations. N Engl J Med. 2020 May 7;382(19):1858-1859. doi: 10.1056/NEJMc2001801. Epub 2020 Apr 6. No abstract available. PMID 32251568
- [Result] Kang H, Kim S, Lee G, Lee I, Lee JP, Lee J, Park H, Moon HB, Park J, Kim S, Choi G, Choi K. Urinary metabolites of dibutyl phthalate and benzophenone-3 are potential chemical risk factors of chronic kidney function markers among healthy women. Environ Int. 2019 Mar;124:354-360. doi: 10.1016/j.envint.2019.01.028. Epub 2019 Jan 17. PMID 30660848
- [Result] Kang H, Lee J, Lee JP, Choi K. Urinary metabolites of organophosphate esters (OPEs) are associated with chronic kidney disease in the general US population, NHANES 2013-2014. Environ Int. 2019 Oct;131:105034. doi: 10.1016/j.envint.2019.105034. Epub 2019 Jul 30. PMID 31374441
- [Result] Lee J, Oh S, Kang H, Kim S, Lee G, Li L, Kim CT, An JN, Oh YK, Lim CS, Kim DK, Kim YS, Choi K, Lee JP. Environment-Wide Association Study of CKD. Clin J Am Soc Nephrol. 2020 Jun 8;15(6):766-775. doi: 10.2215/CJN.06780619. Epub 2020 May 22. PMID 32628126
- [Derived] Kang MW, Kim Y, Lee I, Park H, Park JY, An JN, Yoo KD, Kim YC, Park NY, Kho Y, Choi K, Lee JP, Lee J. Longitudinal behavioral changes and factors related to reinforced risk aversion behavior among patients with chronic kidney disease during the COVID-19 pandemic. Sci Rep. 2022 Sep 22;12(1):15780. doi: 10.1038/s41598-022-19787-0. PMID 36138060